CLINICAL TRIAL: NCT04450628
Title: Esophagogastric Junction Distensibility During Hiatal Hernia Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00081655; 01-20-07 (Other: Atrium); Pro00040539 (Other: Atrium)
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Esophagogastric Junction Distensibility; Hiatal Hernia
Keywords: EndoFLIP; Distensibility of the esophagogastric junction; Gastroesophageal Reflux Disease-Health Related Quality of Life survey; Mayo Dysphagia Questionnaire
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Intervention Model Description: Surgeons will be blinded to EndoFLIP results for half of the cases, with the first 25 cases blinded and the second 25 cases with the surgeons unblinded. There will be interim analysis between the two groups' surgeries. During blinded cases no adjustment will be made to the surgical procedure based on EndoFLIP results, as the operating surgeon will not be informed of the measured values. After the first 25 cases, the surgeons will be unblinded and be able to determine goal impedance planimetry values based on patient postoperative symptom scores.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Surgeons will be blinded to EndoFLIP results for half of the cases, with the first 25 cases blinded and the second 25 cases with the surgeons unblinded. There will be interim analysis between the two groups' surgeries. During blinded cases no adjustment will be made to the surgical procedure based on EndoFLIP results, as the operating surgeon will not be informed of the measured values. After the first 25 cases, the surgeons will be unblinded and be able to determine goal impedance planimetry values based on patient postoperative symptom scores. In the following 25 unblinded cases, the surgeon will be able to augment the surgical intent based on EndoFLIP measurements, such as adding or removing hiatal sutures or repeating the fundoplication . Patients will be blinded to the type of procedure (i.e. surgeon blinded or unblinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgeon blinded (No Intervention): During blinded cases no adjustment will be made to the surgical procedure based on EndoFLIP results, as the operating surgeon will not be informed of the measured values.
  Surgery will be scheduled and patients will undergo intraoperative impedance planimetry with EndoFLIP obtaining measurements of the cross-sectional area, balloon pressure, minimum diameter, compliance, length of high pressure segment, and distensibility index of the EGJ using an 8cm EndoFLIP balloon. Sequential assessments will be performed to 30ml and 40ml for up to a minute for each volume of distension. An initial baseline measurement will be obtained after establishment of pneumoperitoneum. A second measurement will occur following hiatal dissection and mobilization but prior to crural closure. Two additional measurements will be obtained after hiatal closure and after fundoplication.
- Surgeon unblinded (Experimental): The surgeon will be able to augment the surgical intent based on EndoFLIP measurements, such as adding or removing hiatal sutures or repeating the fundoplication. The data will be evaluated to assess if intraoperative calibration influences postoperative symptoms by comparing the two groups.
  Surgery will be scheduled and patients will undergo intraoperative impedance planimetry with EndoFLIP obtaining measurements of the cross-sectional area, balloon pressure, minimum diameter, compliance, length of high pressure segment, and distensibility index of the EGJ using an 8cm EndoFLIP balloon. Sequential assessments will be performed to 30ml and 40ml for up to a minute for each volume of distension. An initial baseline measurement will be obtained after establishment of pneumoperitoneum. A second measurement will occur following hiatal dissection and mobilization but prior to crural closure. Two additional measurements will be obtained after hiatal closure and after fundoplication.
  Interventions: Procedure: Surgeon unblinded; Device: EndoFLIP 1.0 System EF-100

INTERVENTIONS:
Procedure: Surgeon unblinded — The surgeon will be able to augment the surgical intent based on EndoFLIP measurements, such as adding or removing hiatal sutures or repeating the fundoplication. The data will be evaluated to assess if intraoperative calibration influences postoperative symptoms by comparing the two groups.
  Surgery will be scheduled and patients will undergo intraoperative impedance planimetry with EndoFLIP obtaining measurements of the cross-sectional area, balloon pressure, minimum diameter, compliance, length of high pressure segment, and distensibility index of the EGJ using an 8cm EndoFLIP balloon. Sequential assessments will be performed to 30ml and 40ml for up to a minute for each volume of distension. An initial baseline measurement will be obtained after establishment of pneumoperitoneum. A second measurement will occur following hiatal dissection and mobilization but prior to crural closure. Two additional measurements will be obtained after hiatal closure and after fundoplication.
  Other Names: EndoFLIP 1.0 System EF-100
  Arms: Surgeon unblinded
Device: EndoFLIP 1.0 System EF-100 — The surgeon will be able to augment the surgical intent based on EndoFLIP measurements, such as adding or removing hiatal sutures or repeating the fundoplication. The data will be evaluated to assess if intraoperative calibration influences postoperative symptoms by comparing the two groups.
  Surgery will be scheduled and patients will undergo intraoperative impedance planimetry with EndoFLIP obtaining measurements of the cross-sectional area, balloon pressure, minimum diameter, compliance, length of high pressure segment, and distensibility index of the EGJ using an 8cm EndoFLIP balloon. Sequential assessments will be performed to 30ml and 40ml for up to a minute for each volume of distension. An initial baseline measurement will be obtained after establishment of pneumoperitoneum. A second measurement will occur following hiatal dissection and mobilization but prior to crural closure. Two additional measurements will be obtained after hiatal closure and after fundoplication.
  Arms: Surgeon unblinded

SUMMARY:
The investigators aim to ascertain the effects of hiatal hernia repair and fundoplication on the distensibility of the esophagogastric junction (EGJ) as measured by FLIP topography/impedance planimetry. The investigators also aim to assess for any correlation between values of EGJ distensibility and GERD related quality of life (QOL) and dysphagia scores.

DETAILED DESCRIPTION:
Patients referred for antireflux surgery and/or hiatal hernia repair will be considered for enrollment. Standard preoperative evaluation will include esophagogastroduodenoscopy (EGD) to assess for intraluminal pathology including esophagitis, columnar lined esophagus suggestive of Barrett's esophagus, intraluminal masses, and to measure hernia size. Patients will also undergo preoperative high resolution esophageal manometry testing with impedance as clinically indicated to evaluate esophageal motility as assessed by standardized Chicago Classification V3. Manometry will occasionally be avoided in patients with paraesophageal hernias without substantial dysphagia or those not amenable to manometry, with appropriate upper gastrointestinal radiology imaging (UGI), who will be having partial fundoplications. UGI is also a routine preoperative evaluation. Furthermore, pH testing for evaluation of acid reflux will be performed in patients without LA grade C or D esophagitis, paraesophageal hernia, or pathologic confirmation of Barrett's esophagus.

Patients appropriate for enrollment will be consented in the office setting. Preoperative baseline evaluations of symptom severity will be assessed via the GERD-HRQL survey and Mayo Dysphagia Questionnaire. Surgery will be scheduled and patients will undergo intraoperative impedance planimetry with EndoFLIP obtaining measurements of the cross-sectional area, balloon pressure, minimum diameter, compliance, length of high pressure segment, and distensibility index of the EGJ using an 8cm EndoFLIP balloon. Sequential assessments will be performed to 30ml and 40ml for up to a minute for each volume of distension. An initial baseline measurement will be obtained after establishment of pneumoperitoneum. A second measurement will occur following hiatal dissection and mobilization but prior to crural closure. Two additional measurements will be obtained after hiatal closure and after fundoplication.

Surgeons will be blinded to EndoFLIP results for half of the cases, with the first 25 cases blinded and the second 25 cases with the surgeons unblinded. There will be interim analysis between the two groups' surgeries. During blinded cases no adjustment will be made to the surgical procedure based on EndoFLIP results, as the operating surgeon will not be informed of the measured values. After the first 25 cases, the surgeons will be unblinded and be able to determine goal impedance planimetry values based on patient postoperative symptom scores. In the following 25 unblinded cases, the surgeon will be able to augment the surgical intent based on EndoFLIP measurements, such as adding or removing hiatal sutures or repeating the fundoplication. Patients will be blinded to the type of procedure (i.e. surgeon blinded or unblinded). The EndoFLIP catheters and generator will be provided by Medtronic, at no cost to the patient. Medtronic will also cover the fees associated with the EndoFLIP procedure (CPT 91040 is used).

Postoperative clinical care will proceed as per standard protocol for foregut surgery, with 1 additional office visit. Reports of postoperative symptomatology and QOL will be performed, via GERD-HRQL and Mayo Dysphagia Questionnaire during follow up clinic appointments at 2 weeks and 6 weeks postoperative, and with additional long-term follow-up of at 6 months. Long-term follow-up will again assess for QOL symptoms via GERD-HRQL and the Mayo Dysphagia Questionnaire. The 6 month follow-up visit is not typical practice and the patients cost for this visit will be covered by Medtronic. Per standard clinical care, recurrence of symptoms or dysphagia at any point may lead to additional postoperative testing, including UGI, EGD, pH testing, esophageal manometry, CT scan, or EndoFLIP. Postoperative GERD-HRQL and Mayo Dysphagia score results will be compared to intraoperative EndoFLIP measurements in interim and final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing hiatal hernia repair (types I-IV included) and fundoplication
* Absence of spastic esophageal disorders (i.e. jackhammer esophagus, achalasia types I-III) assessed by preoperative high-resolution manometry
* Adult patients ≥18 years
* Elective repairs

Exclusion Criteria:

* Redo hiatal hernia repairs
* Emergent repairs
* Patients with contraindication to surgery or endoscopy
* Patients with esophageal varices
* Cases with insufficient esophageal length in which fundoplication is unable to be performed or a Collis gastroplasty is required
* Connective tissue diseases such as scleroderma or lupus
* Diameter measurements less than 5 mm as the EF-325N catheter is not suitable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in distensibility index | 6 months
  Change in distensibility index of the esophagogastric junction (EGJ) as measured by EndoFLIP before, during, and after hiatal hernia repair (EndoFLIP distensibility index values range from 0 to 98 with higher numbers indicating a tighter EGJ).

SECONDARY OUTCOMES:
Post-op GERD symptoms | 6 months
  Postoperative symptoms as measured by Gastroesophageal Reflux Disease Health Related Quality of Life Questionnaire (GERD-HRQL). The lowest possible score for the GERD-HRQL is 0 and the highest possible score is 75 (higher scores are correlated with worse outcomes).
Post-op dysphagia symptoms | 6 months
  Postoperative symptoms as measured by the Mayo Dysphagia Questionnaire (MDQ-30). The lowest possible score for the MDQ-30 is 0 and the highest score is 100 (higher scores are correlated with worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Colavita, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health - Carolinas Medical Center, Charlotte, North Carolina, United States